CLINICAL TRIAL: NCT00136994
Title: An Open Trial to Evaluate the Efficacy and Tolerability of Ziprasidone IM and Oral in Patients With Psychosis and Acute Agitation.
Brief Title: IM and Oral in Acute Exacerbation of Schizophrenia (BIZET Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1281045
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — ziprasidone

INTERVENTIONS:
Drug: Ziprasidone

SUMMARY:
To evaluate efficacy and tolerability of Ziprasidone IM and oral in agitated patients with acute exacerbation of schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Psychiatric:
* Diagnosis of schizophrenia using DSM-IV (295.xx).
* Patients entering hospital (or inpatients transferring to higher-dependency unit) within the previous seven days because of acute exacerbation of psychotic symptoms.
* PANSS > 80 (score Â³ 3 on at least three of the following PANSS agitation items: anxiety , tension, hostility, excitement).
* CGI-S Â³ 4. - Indication, based on intensity/severity of psychotic symptoms, on IM therapy.
* General:
* Male or Female patients aged 18-60 years at screening.
* Written informed consent to participation.
* Female patients of at risk of pregnancy must avoid to remain pregnant; an adequate method of contraception can be initiated or continued.

Exclusion Criteria:

* Psychiatric:
* Patients at immediate risk of committing harm to self or others
* Concurrent treatment with other antipsychotic agents after baseline
* Patients receiving depot antipsychotic medication within 21 days of screening
* Treatment with antidepressants or mood stabilizers (such as lithium, carbamazepine, valproic acid or verapamil) within two weeks of screening
* Diagnosis of substance abuse using DSM-IV criteria within previous 12 months
* Positive urine drug screen at screening for amphetamine, cocaine or opioids
* Alcohol and/or any other drug abuse at screening
* Patients who have received clozapine within 3 months prior to screening due to intolerance to other antipsychotics or patients who have received clozapine in the past two years for refractoriness to treatment
* Treatment with any investigational agent within the previous six months
* Previous treatment with ziprasidone
* Organic mental disease, including mental retardation
* History of psychosurgery
* General:
* Patients with a history of clinically significant and/or currently relevant hematological, renal (including single kidney), hepatic, gastrointestinal, endocrine (except for current adequately treated hypo- or hyperthyroidism), pulmonary (excluding chronic bronchitis, mild emphysema or chronic obstructive pulmonary disease), dermatological, oncological, or neurological disease, excluding tardive dyskinesia but including all forms of epilepsy (febrile convulsions in childhood acceptable). The only patients with known prior malignant disease who are eligible are those with cured prior skin cancer (excluding melanoma). Controlled Type II diabetes (glucose < 180 mg/100 ml at screening and baseline with dietary or oral hypoglycemic treatment) will not be considered a significant medical illness and would not exclude a subject from the study - Patients with a history of significant cardiovascular disease or significant concurrent cardiovascular disease, including a history of uncontrolled hypertension (supine diastolic pressure >95 mm Hg and/or supine systolic pressure > 170 mm Hg with or without treatment)
* Clinically significant ECG abnormality
* Patient with QTc Â³ 450 msec - Concomitant treatment with medications that prolong QT interval
* Patients with serum K+ or Mg++ outside the normal range
* Confirmed clinically significant laboratory values.
* Known serological evidence of HIV, or acute or chronic hepatitis (with transaminase levels higher than three times the normal limits)
* Patients who intend to donate blood or blood products during the 4 weeks prior to the study, during the study or in the 30 days after the study ends
* Patients unable or unlikely to follow the study protocol
* Pregnant or lactating women
* Patients with a history of neuroleptic malignant syndrome developing from the administration of antipsychotic compounds
* Known hypersensitivity to ziprasidone or lactose

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160
Dates: Start 2003-03; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
To evaluate efficacy and tolerability of Ziprasidone IM and oral in agitated patients with acute exacerbation of schizophrenia

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- Italy (33):
  - Pfizer Investigational Site, Savigliano, Cuneo
  - Pfizer Investigational Site, Campi Bisenzio, Firenze
  - Pfizer Investigational Site, Sora, Frosinone
  - Pfizer Investigational Site, Parma, PR
  - Pfizer Investigational Site, S. Arsenio, Salerno
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Cagliari
  - Pfizer Investigational Site, Caserta
  - Pfizer Investigational Site, Chiari (BS)
  - Pfizer Investigational Site, Cremona
  - Pfizer Investigational Site, Fidenza(pr)
  - Pfizer Investigational Site, Foggia
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Genova-sestri
  - Pfizer Investigational Site, Lecce
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Modena
  - Pfizer Investigational Site, Moncalieri(to)
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Noto
  - Pfizer Investigational Site, Orbassano (TO)
  - Pfizer Investigational Site, Padua
  - Pfizer Investigational Site, Palermo
  - Pfizer Investigational Site, Perugia
  - Pfizer Investigational Site, Pordenone
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Sassari
  - Pfizer Investigational Site, Senigallia (AN)
  - Pfizer Investigational Site, Torino
  - Pfizer Investigational Site, Torrette DI Ancona (AN)
  - Pfizer Investigational Site, Udine
  - Pfizer Investigational Site, Verona
  - Pfizer Investigational Site, Viareggio